CLINICAL TRIAL: NCT03748914
Title: The Influence of Cut-umbilical Cord Milking (C-UCM) on the Cerebral Oxygenation and Perfusion of Preterm and Term Infants
Brief Title: C-UCM and Cerebral Oxygenation and Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 30-450 ex 17/18; U1111-1223-3280 (Other: WHO Universal Trial Number (UTN))
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Preterm Infant; Term Infant; Transition
MeSH Terms: conditions — Premature Birth | interventions — Control Groups; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Milking the cut umbilical cord once towards the Infant at a speed of 10cm/second.
  Interventions: Other: Intervention Group
- Control Group (Active Comparator): The umbilical cord is cut according to the standard procedure and no C-UCM is performed.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Group — After delivery of the neonate via caesarean section the umbilical cord will be clamped within 30 seconds and cut long at least 30 cm by the obstetrician. The neonate is then placed under an overhead heater by the midwife. There, the umbilical cord must be untwisted and held in a vertical position. It is milked once by the neonatologist towards the baby at a speed of approximately 10 cm/s and then clamped 3 cm from the umbilicus by one member of the clinical team.
  Other Names: Cut umbilical cord milking (C-UCM)
  Arms: Intervention Group
Other: Control Group — The umbilical cord is cut according to the standard procedure and no C-UCM is performed.
  Other Names: Standard care
  Arms: Control Group

SUMMARY:
In this randomized controlled Pilot study the effects of cut-umbilical cord milking on cerebral oxygenation and perfusion measured via near-infrared spectroscopy (NIRS) and the effects on stroke volume (SV) and cardiac output (CO) also measured non-invasively in term and preterm infants are evaluated for the first 15 minutes after birth and compared to a control group.

DETAILED DESCRIPTION:
Background

The transition to life after birth is a complex physiological process where the neonate has to establish sufficient ventilation and changes from intra-uterine circulation to extra-uterine circulation take place. During these processes the neonate has to provide the brain with adequate perfusion and oxygen delivery to maintain normal cerebral tissue oxygenation and activity. Instability of cerebral perfusion and oxygenation may be associated with brain damage in preterm infants. The concept of C-UCM may substitute the adverse effects of immediate cord clamping by supplying additional placental blood to the infant, which is mostly performed during caesarean section or in the critically ill neonate.

In this randomized controlled Pilot study the effects of cut-umbilical cord milking on cerebral oxygenation and perfusion measured via near-infrared spectroscopy (NIRS) and the effects on stroke volume (SV) and cardiac output (CO) also measured non-invasively in term and preterm infants are evaluated for the first 15 minutes after birth and compared to a control group.

Aim

The aim of the study is to analyse whether C-UCM in preterm and term infants results in an improvement of cerebral oxygenation and perfusion during immediate neonatal transition measured with NIRS.

Hypotheses

Infants undergoing C-UCM after birth compared to infants without C-UCM show differences in cerebral oxygenation and perfusion in the first 15 min after birth.

Hypothesis I: C-UCM and cerebral blood volume (CBV) In infants with C-UCM there is more CBV decrease immediately after birth, compared to infants without C-UCM, due to improved cerebral oxygen delivery.

Hypothesis II: C-UCM and cerebral regional oxygen saturation (crSO2) Infants with C-UCM have higher crSO2 values during immediate neonatal transition, compared to infants without C-UCM, again due to improved cerebral oxygen delivery.

Hypothesis III: C-UCM and stroke volume (SV) In infants with C-UCM the SV at 15 minutes after birth is higher, compared to infants without C-UCM

Hypothesis IV: C-UCM and cardiac output (CO) In infants with C-UCM the CO at 15 minutes after birth is higher, compared to infants without C-UCM.

Hypothesis V: C-UCM and mean arterial blood pressure (MABP) In infants with C-UCM the MABP at 5, 10 and 15 minutes after birth is higher, compared to infants without C-UCM.

Study population

Preterm infants Neonates with a gestational age ≥28 - 37 weeks delivered by caesarean section at the Department of Obstetrics and Gynaecology, Medical University of Graz, will be enrolled into the study, provided written informed consent is obtained from parents prior to birth. Neonates with severe congenital malformations will be excluded.

Term Infants Neonates with a gestational age ≥37 weeks delivered by caesarean section at the Department of Obstetrics and Gynaecology, Medical University of Graz, will be enrolled into the study, provided written informed consent is obtained from parents prior to birth. Neonates with severe congenital malformations will be excluded.

Study design

The present study is designed as a randomized controlled pilot trial. As there have not been prior human studies investigating C-UCM regarding the outcome measures cerebral oxygenation and perfusion, a randomized controlled pilot study is the appropriate first step to be able to calculate sample size for a bigger trial.

Sample Size

Sample size calculations were not performed, since there are no data from previous human studies available, and this pilot study needs to be conducted to generate data for the sample size calculation of a consecutive main study. For this pilot study a sample size of 80 infants (20 subjects in the intervention group of preterm infants, 20 subjects in the intervention group of term infants, 20 subjects in each of the two control groups) is arbitrary designated.

Procedure

The medical history focussing on any pathologic findings during pregnancy and delivery will be collected and stored anonymously.

After delivery of the neonate via caesarean section, in the intervention group the umbilical cord will be clamped within 30 seconds and cut long at least 30 cm by the obstetrician. The neonate is then placed under an overhead heater by the midwife. There, the umbilical cord must be untwisted and held in a vertical position. It is milked once by the neonatologist towards the baby at a speed of approximately 10 cm/s and then clamped 3 cm from the umbilicus by one member of the clinical team. In contrast, in the control group the umbilical cord is cut according to the standard procedure and no C-UCM is performed. The further treatment procedure is the same in both groups.

A NIRS transducer will be placed on the newborn's left forehead, and fixed with a modified neonatal CPAP cap or gauze bandage by a scientific staff member without disturbing routine medical care. Furthermore, a pulse oximeter sensor will be attached on the right wrist or palm to monitor preductal oxygen saturation by pulse oximetry (SpO2) and heart rate (HR). Moreover 4 electrodes are fixed on the skin for the non-invasive cardiac output monitoring (NICOM) to evaluate SV and CO. All the measurements will be performed within the first 15 minutes after birth.

Intervention The pneumatic cuff for the oscillometric measurements of the arterial blood pressure will be placed around the left upper arm (or alternatively on the left lower leg) at 5, 10 and 15 minutes after birth. A capillary blood gas check 15 minutes after birth will be performed in all the patients; However infants in need for respiratory support during postnatal stabilisation receive this blood gas check routinely. Moreover, rectal temperature will be measured at 15 minutes after birth.

A stopwatch is started at delivery, the time points of umbilical cord clamping, C-UCM in the intervention group, establishment of NIRS measurement, establishment of SpO2 measurement, and blood drawing for the gas check will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with a gestational age ≥28 weeks
* Delivered by caesarean section
* Decision to conduct full life support
* Written informed consent prior to birth

Exclusion Criteria:

* Neonates with a gestational age <28 weeks
* No decision to conduct full life support
* No written informed consent
* Severe congenital malformations

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Cerebral blood volume | within the first 15 minutes after birth.
  Changes in CBV (ml/100g brain)

SECONDARY OUTCOMES:
Cerebral tissue oxygenation index | within the first 15 minutes after birth
  Changes in cTOI (%)
Peripheral oxygen saturation | within the first 15 minutes after birth
  Changes in SpO2 (%)
Heart rate | within the first 15 minutes after birth
  Changes in HR (beats per minute)
Stroke volume | within the first 15 minutes after birth
  Changes in SV (ml)
Cardiac output | within the first 15 minutes after birth
  Changes in CO (l/min)
Mean arterial blood pressure | within the first 15 minutes after birth
  Changes in MABP (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Berndt Urlesberger, Professor, Principal Investigator — Division of Neonatology, Medical University of Graz
Locations (1):
- Dep. of Pediatrics, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/14/NCT03748914/Prot_SAP_000.pdf